CLINICAL TRIAL: NCT02163928
Title: Evaluation of Changes in Skin Carotenoid Scores in Medical Students Following Dietary Interventions
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L14-128; CRI14-042 Skin Carotenoids (Other: Clinical Research Institute)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Health Behavior
Keywords: Antioxidants; Carotenoids; Diet
MeSH Terms: conditions — Health Behavior | interventions — Vegetables

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Food-based intervention; increased fruits and vegetables — 4-6 cups of fruits and vegetables daily for 8-weeks
  Other Names: Whole-diet intervention

SUMMARY:
Skin Carotenoid Scores (SCS) are a biomarker of overall antioxidant status. This study will use Raman Spectroscopy to examine the ability of increased dietary intake of fruits and vegetables to increase SCS in medical students. This will be an observational, non-invasive study examining skin carotenoid levels over time in individuals who have increased their intake by dietary adjustments. Thirty medical students meeting study inclusion criteria will be asked to increase their intake of high antioxidant fruits and vegetables to 4-6 cups per day over an eight week period of time. Students will self-select their fruits and vegetables from a given list and will receive supermarket gift cards to offset the cost of the increased food. Students will be asked to follow their usual diet for one week. Then increase their intake of high antioxidant fruit and vegetable to 4-6 cups per day for eight weeks. Then return to their usual diet for 2 weeks. SCS scores will be taken at baseline and week 1. At the beginning of week 2, students will be asked to increase fruit and vegetable intake to 4-6 cups per day. SCS will be measured every two weeks during the 8-week intervention phase. Students will return to their usual diet for 2 weeks and SCS will be measured at the end of that 2-week period.

DETAILED DESCRIPTION:
Inclusion criteria:

* Medical students (any year) from Texas Tech School of Medicine
* BMI between 20-29
* Non-smoker, non-pregnant

Exclusion criteria:

* Individuals suffering from a chronic disease such as diabetes, heart disease, or other metabolic disorder
* Pregnant women
* Smokers
* Individuals with BMI > or = 30 or < or = 19

ELIGIBILITY:
Inclusion Criteria:

* Medical student from any year at Texas Tech University School of Medicine willing to maintain the increased consumption of fruits and vegetables for the entire eight-week experimental period, to maintain logs and to report at each of the times that measurements will be taken.

Exclusion Criteria:

* Pregnancy
* Smoker
* BMI =/> 30
* Chronic disease such as diabetes, heart disease, or metabolic disorder

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical students from Texas Tech University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Skin Carotenoid Scores (SCS) | Baseline, 2,4,6,8,10,12 weeks
  Skin Carotenoid Scores (SCS) are a biomarker of overall antioxidant status. The purpose of this study is to measure changes in SCS in medical students when fruit and vegetable consumption is increased. SCS will measured using a Bio-photonic Scanner. This scanner non-invasively measures carotenoid levels in the skin using optical signals. By placing the palm of the hand in front of a low-energy blue light for less than two minutes, the scanner can determine the SCS.

SECONDARY OUTCOMES:
Body weight | Baseline, 2,4,6,8,10,12 weeks
  Weight will be measured on a calibrated balance scale. Subjects will remove shoes, keys, cellphones, or other objects from their person before being weighed.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Chauncey, PhD, RDN, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

REFERENCES:
- [Background] Ermakov IV, Ermakova MR, McClane RW, Gellermann W. Resonance Raman detection of carotenoid antioxidants in living human tissues. Opt Lett. 2001 Aug 1;26(15):1179-81. doi: 10.1364/ol.26.001179. PMID 18049555
- [Background] Ermakov IV, Gellermann W. Validation model for Raman based skin carotenoid detection. Arch Biochem Biophys. 2010 Dec 1;504(1):40-9. doi: 10.1016/j.abb.2010.07.023. Epub 2010 Aug 1. PMID 20678465
- [Background] Mayne ST, Cartmel B, Scarmo S, Lin H, Leffell DJ, Welch E, Ermakov I, Bhosale P, Bernstein PS, Gellermann W. Noninvasive assessment of dermal carotenoids as a biomarker of fruit and vegetable intake. Am J Clin Nutr. 2010 Oct;92(4):794-800. doi: 10.3945/ajcn.2010.29707. Epub 2010 Aug 4. PMID 20685953
- [Background] Mayne ST, Cartmel B, Scarmo S, Jahns L, Ermakov IV, Gellermann W. Resonance Raman spectroscopic evaluation of skin carotenoids as a biomarker of carotenoid status for human studies. Arch Biochem Biophys. 2013 Nov 15;539(2):163-70. doi: 10.1016/j.abb.2013.06.007. Epub 2013 Jun 30. PMID 23823930
- [Background] Meinke MC, Darvin ME, Vollert H, Lademann J. Bioavailability of natural carotenoids in human skin compared to blood. Eur J Pharm Biopharm. 2010 Oct;76(2):269-74. doi: 10.1016/j.ejpb.2010.06.004. Epub 2010 Jun 15. PMID 20558286